CLINICAL TRIAL: NCT03833947
Title: Comparision of Addition of Dexamethasone vs Bicarbonate to Intracuff Lignocaine 2% in Terms of Extubation Characteristics and Patient Satisfaction Undergoing General Anaesthesia
Brief Title: Dexamethasone vs Bicarbonate to Intracuff Lignocaine 2% in General Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aligarh Muslim University (Other)
Responsible Party: Principal Investigator, MUAZZAM HASAN, Assistant Professor, Department of Anaesthesiology, Aligarh Muslim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AligarhMUmzm
Record Dates: First submitted 2019-01-24; First posted 2019-02-07 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia; Anesthesia; Adverse Effect; Anesthesia Intubation Complication
Keywords: Intracuff Dexamethasone; Intracuff Alkalinized lignocaine; General anesthesia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lignocaine with bicarbonate (Experimental): Endotracheal tube cuff was filled with mixture of 7.5% sodium bicarbonate with 2% lignocaine in a ratio of 0.5:9.5 ml
  Interventions: Drug: lignocaine+bicarbonate
- lignocaine with dexamethasone (Active Comparator): Endotracheal tube cuff was filled with mixture of dexamethasone with 2% lignocaine in a ratio of 0.5:9.5 ml
  Interventions: Drug: lignocaine+dexamethasone

INTERVENTIONS:
Drug: lignocaine+bicarbonate — ETT cuff was filled with mixture of 2% lignocaine with bicarbonate
  Arms: lignocaine with bicarbonate
Drug: lignocaine+dexamethasone — ETT cuff was filled with mixture of 2% lignocaine with dexamethasone
  Arms: lignocaine with dexamethasone

SUMMARY:
This study is designed to evaluate and compare the effect on hemodynamics, extubation response and patients satisfaction score in patients with ETT cuff filled with either mixture of lignocaine with sodium bicarbonate or with a mixture of lignocaine with dexamethasone.

DETAILED DESCRIPTION:
Objective Recently multiple studies have shown better outcomes with usage of dexamethasone or alkalinized lignocaine instead of air for filling endotracheal tube (ETT) cuff. So this study is designed to evaluate and compare the effect on hemodynamics, extubation response and patients satisfaction score in patients with ETT cuff filled with either mixture of lignocaine with sodium bicarbonate or with a mixture of lignocaine with dexamethasone.

Design and setting:

This is a prospective single blind, randomized controlled study at the department of anesthesiology, JNMCH, AMU, Aligarh.

Materials and methods:

Investigators plan to include 100 patients of age group within 18-60 years with American Society of Anesthesiologists (ASA) class I & II, posted for elective surgery of duration >120 minutes, performed under general anesthesia; administered as per institutional protocols. Patients with ASA III & IV, cardiovascular morbidities, known drug allergy, pregnancy will be excluded from the study. Patients will be divided into two groups randomly according to chit-in-box method, viz Group A & Group D with fifty patients in each group. Patient group allocation, preparation of drug mixture for endotracheal cuff filling as per group assigned and analysis of observed data will be done by a separate anesthetist not involved in the perioperative management of the patient. In patients belonging to Group (A), ETT cuff will be filled with mixture of 7.5% sodium bicarbonate with 2% lignocaine in the proportions of 0.5: 9.5 ml while in Group D the ETT cuff will be filled with mixture of dexamethasone with 2% lignocaine in the proportions of 0.5: 9.5 ml . The cuff of the ETT will be slowly inflated until no leak is heard at all during the peak airway pressure of the ventilator cycle while auscultating the trachea . Volume of drug mixture in the cuff will be noted at start and end of surgery. Total duration of anesthesia will be noted.

Hemodynamic stability at the time of extubation will be meausred in terms of changes in rate pressure product (RPP) which will denote the product of heart rate and systolic blood pressure. RPP values recorded immediately after stoppage of the anesthetic agents at the end of surgery will be compared to the values measured just after the extubation of trachea. Patient's satisfaction from anesthesia given will be recorded, based on VAS. The presence of coughing and bucking will also be noted. Incidence of postoperative sore throat and cough will be recorded at 1 hour and 24 hours post extubation.

The results will be presented in number, percentage, mean, and standard deviation as appropriate. Appropriate statistical tests will be applied and P value less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I & II.
* Elective surgery
* General anesthesia of duration >120 minutes.

Exclusion Criteria:

* Patients with ASA III & IV.
* Known Cardiovascular morbidities.
* Pregnancy.
* Allergic to used drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
smoothness of extubation | time from adequate reversal of anaesthesia & muscle paralysis (head holding >5sec, eye opening on command, train of four ratio >0.9) till removal of endotracheal tube.
  Grade 1= coughing, bucking, tube biting, agitatation present. Grade 2= mild bucking/coughing. Grade 3= completely comfortable, tolerating tube in situ, no coughing/bucking/agitation.
patient satisfaction score | post operative 1 hour
  rated on visual analog scale varying 0 to 10; where 0 is worst experience and 10 is best. completely

SECONDARY OUTCOMES:
Haemodynamic stability at the time of extubation. | values of product of systolic blood pressure and heart rate will be compared after stopping the anesthetic agents and immediately after the extubation
  Rate pressure product (RPP); [RPP=Product of systolic blood pressure(mmHg) and heart rate (beats per min)] measured after stopping the anaesthetic agents at the end of surgery will be taken as baseline and then compared to values measured immediately after the removal of endotracheal tube.
amount of drug diffused through endotracheal tube cuff | from start till end of surgery.
  Volume of drug mixture in the cuff was noted at start and end of surgery.
incidence of post operative cough and sore throat | after 1 and 24 hour post extubation
  incidence of post operative cough and sore throat

OTHER OUTCOMES:
duration of surgery | duration of surgery
  duration of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Jawaharlal Nehru Medical College, Aligarh, Uttar Pradesh, India